CLINICAL TRIAL: NCT00654888
Title: Study of Automated Lamellar Keratectomy With a New Option in Treatment in Symptomatic Patients With Bullous Keratopathy.
Brief Title: Automated Lamellar Keratectomy in Symptomatic Patients With Bullous Keratopathy
Acronym: ALKSBK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Eliana Domingues Gonçalves, UNIFESP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0068/05
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Corneal Disease
Keywords: cataract extraction; surgery; corneal disease
MeSH Terms: conditions — Corneal Diseases | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Group one submitted to automated lamellar keratectomy(ALK) with mitomycin (0,02% in 30 seconds after keratectomy).
  Interventions: Drug: Mitomycin
- 2 (Active Comparator): automated lamellar keratectomy without mitomycin
  Interventions: Procedure: ALK (automated lamellar keratectomy)

INTERVENTIONS:
Procedure: ALK (automated lamellar keratectomy) — ALK is performed with a microkeratome, to make a free cap.
  Other Names: automated lamellar keratectomy with PTK
  Arms: 2
Drug: Mitomycin — mitomycin 0,02%, 30 seconds after ALK
  Other Names: automated lamellar keratectomy associated with PTK
  Arms: 1

SUMMARY:
To relieve pain in patients with symptomatic bullous keratopathy (BK) until keratoplasty and in patients without visual prediction.

The automated lamellar keratectomy represents a alternative in treatment of pain in symptomatic patients with BK.

DETAILED DESCRIPTION:
Only patients with BK symptomatic (with pain) were submitted to automated lamellar keratectomy (ALK).

Complete ophthalmological examination including UCVA,BSVA, biomicroscopy, tonometry, esthesiometry, UBM pachymetry, impression cytology and pain questionnaire were performed in preoperative, postoperative of one, seven, 30, 90, 180 days and one year.

ELIGIBILITY:
Inclusion Criteria:

* Patient with bullous keratopathy symptomatic (with pain)

Exclusion Criteria:

* herpetic endotelial disorders

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pain questionnaire | preoperative and postoperative 1,7,30,90,180 days and one year

SECONDARY OUTCOMES:
biomicroscopy, esthesiometry, UBM pachymetry, impression cytology | preoperative, postoperative 1,7,30,90,180 days and one year

CONTACTS AND LOCATIONS:
Overall Officials: Eliana D Gonçalves, MD, Principal Investigator — Federal University of São Paulo